CLINICAL TRIAL: NCT02134431
Title: Dose-response Relationship of Tenofovir With HIV-1 Suppression in ex Vivo Model of Tissue Infectibility in Adolescents
Brief Title: Relationship of Tenofovir With HIV-1 Suppression in ex Vivo Tissue in Adolescents
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: UL1TR000124-1955; UL1TR000124 (NIH)
Record Dates: First submitted 2014-05-02; First posted 2014-05-09 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; tenofovir; miocrobicide; endoscopy (colonoscopy, sigmoidoscopy); adolescents; pediatrics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Colonoscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV positive: HIV-positive subjects ages 10-14 years old and 18-21 years old taking tenofovir in their antiretroviral regimen.HIV positive subjects will undergo lower endoscopy (specifically either flexible sigmoidoscopy or colonoscopy) with biopsies to obtain colorectal tissue samples. HIV-1 levels and tenofovir levels in tissue will be measured.
  Interventions: Device: flexible sigmoidoscopy or colonoscopy with biopsies
- HIV negative: HIV-negative subjects ages 10-14 years old and 18-21 years old. HIV negative subjects will undergo lower endoscopy (specifically either flexible sigmoidoscopy or colonoscopy) with biopsies to obtain colorectal tissue samples. These tissue samples will be pretreated with tenofovir and challenged with laboratory HIV-1.
  Interventions: Device: flexible sigmoidoscopy or colonoscopy with biopsies

INTERVENTIONS:
Device: flexible sigmoidoscopy or colonoscopy with biopsies — Lower endoscopy with biopsies (specifically either colonoscopy or flexible sigmoidoscopy) in both HIV-positive subjects already on oral tenofovir , as well as HIV negative subjects. Biopsies will be taken to laboratory for quantification of HIV-1 and drug levels of tenofovir.

SUMMARY:
Microbicides are topical medicines that can prevent infection by Human Immunodeficiency Virus (HIV). Microbicide medicine has yet to be studied in adolescents, a key group that is becoming infected with HIV all over the world. From past research, we know that at different ages people experience age-related changes in their bodies that can cause differences in how they process medications. In this study, gut tissue samples (or gut biopsies) from 12 HIV-negative volunteers will be collected. These pieces of tissue will be infected with HIV in the laboratory to develop a model that can be used to test certain drugs against the HIV infection. We can use this tissue to test a drug called tenofovir against HIV infection. We will determine whether this drug can decrease HIV infection in the gut biopsies. In this study, we will also measure HIV levels and the levels of tenofovir in gut and blood samples in 12 people who are already taking this drug. This information can determine whether levels of drug found in the gut can protect it from HIV. The results can be compared to other age groups of adolescents and adults. Subjects will undergo a common procedure called a lower endoscopy (this can be a colonoscopy or a flexible sigmoidoscopy) to obtain gut biopsy samples.

The central hypothesis is that tissue drug profiles of tenofovir (TFV) and its active component, tenofovir disoproxil fumarate (TDF), and tissue infectibility vary between younger (10-14 years old) versus older adolescents (18-21 years old), and that both differ from adults (>21 years). Specifically, younger HIV positive adolescents will have lower levels of tissue tenofovir compared to older HIV positive adolescents and adults in an age-dependent manner. Additionally, biopsies from younger HIV negative adolescents will have: 1) higher rates of infection compared to biopsies from older HIV negative adolescents infected with a lower dose of virus; and 2) lower percent suppression of tissue infectivity compared to biopsies from older HIV negative adolescents using low dose tenofovir.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 10 years and </= 14 years and age </= 18 years and </= 21 years.
2. Willing and able to communicate in English.
3. Willing and able to provide written informed consent or assent to take part in the study (where required, parent/guardian must provide consent).
4. Willing and able to provide adequate information for locator purposes.
5. Understand and agree to local sexually transmitted infections (STI) reporting requirements.
6. HIV-negative or -positive as documented in prior serologic testing or per report, and willing to undergo repeat HIV testing.
7. Willing and able to not take aspirin, any aspirin containing medications, or non-steroidal anti-inflammatory drugs for at least 72 hours before and 72 hours after flexible sigmoidoscopy.
8. All female patients of childbearing potential (post-menarche) must be willing to undergo urine pregnancy testing at screening.
9. Must be in general good health, including normal renal function.
10. Subjects <18 years old must be scheduled for a clinically indicated colonoscopy or flexible sigmoidoscopy with biopsies.
11. HIV-positive participants only (Aim 1):

    * Must have recent HIV polymerase chain reaction (PCR) documented in the last 6-12 months by verbal report
    * Must have tenofovir in chronic cART regimen (>/= 1 month).
    * Be reportedly compliant.
    * CD4 T cells >250/cmm

Exclusion Criteria:

1. Known history of inflammatory bowel disease.
2. Abnormalities of the colorectal mucosa, or significant colorectal symptom(s) which in the opinion of the clinician represents a contraindication to biopsy (including but not limited to presence of any unresolved injury, inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids).
3. Evidence of any known enteric infection at the time of study visit.
4. Participant-reported symptoms and/or clinical or laboratory diagnosis of active and symptomatic rectal infection (gonorrhea, Chlamydia, syphilis, clinically active perineal HSV).

   * Note: Allow one re-screening after documented treatment (30 days) in cases of gonorrhea/chlamydia (GC/CT) identified at screening.
5. Pregnancy.
6. Subjects with other poorly controlled medical conditions (e.g. diabetes, congestive heart failure).
7. Chronic renal disease (BUN and serum creatinine >1.5 times the upper normal limit).
8. History or presence of impaired gastrointestinal motility, or history of extensive small bowel resection (greater than half the length of the small intestine).
9. Use of warfarin or heparin.
10. Use of systemic immunomodulatory medications within 4 weeks of screening.
11. Use of any investigational products within 4 weeks of screening.
12. Fever at time of endoscopy. Subjects can be re-scheduled at a later point after the fever is resolved.
13. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of sever, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: HIV positive adolescents already taking tenofovir in their antiretroviral regimen. Must be 10-14 years (n=6) and 18-21 years (n=6). HIV negative adolescents who are otherwise healthy ages10-14 years (n=6) and 18-21 years (n=6). Recruitment will be voluntary from the city/community and outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measure Cmax of tenofovir (TFV) in plasma (ng/ml) & tissue (ng/mg), tenofovir-diphosphate (TFV-DP) in tissue (fmol/mg) and PBMC (fmol/million), HIV quantified PCR (copies/ml) from tissue & plasma. | 1 year
  Quantification of TFV and TFV-DP drug concentrations by LC-MS/MS (Liquid chromatography-mass spectrometry/mass spectrometry), and HIV-1 viral load in colorectal biopsies, plasma, and peripheral blood mononucleated cell (PBMC) of HIV positive adolescents.
  Measure TFV in plasma (ng/ml) and tissue (ng/mg). Measure TFV-DP in tissue (fmol/mg) and PBMC (fmol/million). Measure HIV quantified PCR (copies/ml) from colorectal biopsy tissues and plasma.
establish ex vivo infectibility assay as measured by HIV-1 p24 (pg/ml) in HIV-negative biopsies infected with R5 HIV-1BaL low 10^2 TCID50 or high 10^4 TCID50 concentration | 1 year
  After infecting gut biopsy samples ex vivo from HIV negative subjects with either low (10^2 TCID50 ) or high (10^4 TCID50) titer of R5 HIV-BaL), supernatants will collected every 3-4 days for HIV-1 p24 (pg/ml) quantification by ELISA. This quantification will assess viral replication in biopsy tissues.
Assess differences in percent suppression of tissue infectivity (measured by HIV-1 p24 (pg/ml)) in biopsies from younger vs older adolescents pretreated with low dose tenofovir. | 1 year
  Mucosal biopsies will be pretreated with low-dose tenofovir ex vivo. Pretreated biopsies will then be infected with either 10^2 TCID50 or 10^4 TCID50 R5 HIV-1BaL. Supernatants will be collected every 3-4 days over a 14 day period for HIV-1 p24 (pg/ml) by ELISA. Percent suppression of tissue infectivity in biopsies will be assessed and compared between age groups.

SECONDARY OUTCOMES:
Measures of tenofovir drug efficacy predicting drug levels (tissue TFV ng/mg, TFV-DP fmol/mg) necessary to suppress 50%, 90%, 95% of biopsy HIV-1 p24 (pg/ml) (EC50,90,95) will be calculated by interpolation of the dose response curve. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sue McDiarmid, MD, Principal Investigator — University of California, Los Angeles, Departments of Pediatrics and Surgery
Locations (1):
- UCLA Clinical and Translational Research Center (CTRC), Los Angeles, California, United States